CLINICAL TRIAL: NCT00882557
Title: A Prospective, Randomized, Crossover-design Study to Evaluate the Pharmacokinetics and Safety of Daptomycin Administered at 9 mg/kg During and 6 mg/kg After Hemodialysis
Brief Title: Study to Evaluate Daptomycin Given During Dialysis and After Dialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3009-027; DAP-RENID-08-06 (Other: Cubist Study Number)
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Results first posted 2011-10-25 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-01

CONDITIONS: End-stage Renal Disease; Renal Failure Chronic Requiring Hemodialysis
Keywords: End-stage renal disease; hemodialysis; chronic renal failure
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Daptomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): 9 mg/kg of daptomycin administered during the last 30 minutes of a hemodialysis session.
  Interventions: Drug: daptomycin
- B (Experimental): Post dialysis dosing
  Interventions: Drug: daptomycin

INTERVENTIONS:
Drug: daptomycin — intradialytic: 9 mg/kg during the last 30 minutes of dialysis
  Other Names: Cubicin
  Arms: A
Drug: daptomycin — 6 mg/kg administered after a hemodialysis session
  Other Names: Cubicin
  Arms: B

SUMMARY:
The purpose of this study is to determine whether daptomycin at a higher dose given during the last 30 minutes of a dialysis session is equal to a lower dose of daptomycin given after a dialysis session.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to any study-related procedure not part of normal medical care;
* Male or female ≥ 18 years of age;
* If female of childbearing potential; willing to practice reliable birth control measures during study treatment and for at least 28 days after study completion, not lactating or pregnant, and has a documented negative pregnancy test result within 24 hours prior to study medication administration;
* End-stage renal disease on stable (for at least 2 weeks) hemodialysis regimen, three times weekly using high-flux membranes;
* Functioning hemodialysis access (for example, graft or fistula);
* Considered to be in appropriate health for study entry by the Investigator (for example, no acute, debilitating medical problems) and appropriate candidate for completing study treatment;
* If taking concomitant medications, subject must be on a relatively stable dose for at least two weeks prior to study drug administration.

Exclusion Criteria:

* Received an investigational drug (including experimental biologic agents) within 30 days of study drug administration;
* Has received any dose of daptomycin within 7 days prior to study drug administration;
* Known to be allergic or intolerant to daptomycin;
* Evidence of active ongoing infection;
* Known human immunodeficiency virus (HIV) infection with CD4 count ≤ 200 cells/mm3;
* Active illicit drug use or alcohol abuse;
* Myocardial infarction within last 6 months;
* Subject with a history of muscular disease (for example, polymyositis, muscular dystrophy);
* Subject with a history of neurological disease (for example, Guillain Barré, multiple sclerosis), except stroke > 6 months prior to study entry;
* Intramuscular injection within 7 days of study drug administration;
* Body mass index (BMI) ≤ 18.5 or ≥ 40 kg/m2 (BMI = weight [kg]/height [m2]);
* WBC ≥ 12, 000 cells/mm3 or ≤ 2500 cells/ mm3;
* Neutropenic subject with absolute neutrophil count ≤ 500 cells/mm3;
* Baseline CPK values ≥ 3X ULN (upper limit of normal);
* Alanine aminotransferase (ALT) > 5XULN;
* Aspartate aminotransferase (AST) > 5XULN;
* Hemoglobin ≤ 9 gm/dL;
* Is considered unlikely to comply with study procedures or to return for scheduled post-treatment evaluations;
* History of rhabdomyolysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-04-29 (Actual); Primary Completion 2009-07-17 (Actual); Study Completion 2009-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alistair Wheeler, MD, MFPM, Study Director — Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)
Locations (2):
- United States (2):
  - West Coast Clinical Trials, Cypress, California
  - DaVita Clinical Research, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects evaluated for entry within 7 days prior to randomization, washout period of 7-14 days between doses, subjects began Day 1 on Friday of Monday/Wednesday/Friday or Saturday of Tuesday/Thursday/Saturday hemodialysis schedule
Groups:
- Sequence BA: All subjects received 1 dose of daptomycin 6 mg/kg after hemodialysis (Regimen B) and 1 dose of daptomycin 9 mg/kg during the last 30 minutes of hemodialysis (Regimen A).
- Sequence AB: All subjects received 1 dose of daptomycin 9 mg/kg during the last 30 minutes of hemodialysis (Regimen A) and 1 dose of daptomycin 6 mg/kg after hemodialysis (Regimen B).
Period: Overall Study
Arm/Group | Sequence BA | Sequence AB
Started | 8 | 8
Completed Dose 1 | 8 | 7
Completed Dose 2 | 6 | 7
Completed | 6 | 7
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Trouble with Vein Access | 1 | 0
Not completed — Randomized Not Treated | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence BA | Sequence AB | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] — Safety population (1 patient included in the overall number of baseline participants in the "Sequence AB" arm was randomized but not treated)
  years | 51.6 (13.19) | 55.3 (6.05) | 53.3 (10.31)
Sex: Female, Male [Count of Participants; unit: Participants] — Safety population (1 patient included in the overall number of baseline participants in the "Sequence AB" arm was randomized but not treated)
  Participants
    Female | 3 | 1 | 4
    Male | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Area Under the Curve From Time 0 to Infinity
Description: Area under the plasma concentration versus time curve from time 0 to infinity for daptomycin doses
Time Frame: Within 30 minutes prior to the start of the infusion, mid-infusion, and end of the infusion; at 1, 2, 4, 6, 9, 24, and 48 hours after the end of the infusion; and just prior to the next hemodialysis session (i.e., 68 hours post-infusion)
Population: The primary endpoints are measured on the PK population, defined as all subjects who received both the 6 mg/kg dose and 9 mg/kg dose
Measure: Median (Full Range); unit: hr*ug/mL
Groups:
- 6 mg/kg After Hemodialysis (Regimen B): Daptomycin (6 mg/kg IV) after hemodialysis using high-flux membranes
- 9 mg/kg During Hemodialysis (Regimen A): Daptomycin (9 mg/kg IV) during the last 30 minutes of hemodialysis using high-flux membrane
Arm/Group | 6 mg/kg After Hemodialysis (Regimen B) | 9 mg/kg During Hemodialysis (Regimen A)
Number analyzed (Participants) | 13 | 13
hr*ug/mL | 1692 [962 to 2524] | 2708 [1719 to 4010]

2. Other Pre Specified Outcome: Maximum Plasma Concentration
Description: Maximum plasma concentration over the entire sampling phase directly obtained from the experimental plasma concentration time data, without interpolation.
Time Frame: as for outcome 1
Population: PK Population - defined as all subjects who received both doses of daptomycin
Measure: Median (Full Range); unit: ug/mL
Arm/Group | 6 mg/kg After Hemodialysis (Regimen B) | 9 mg/kg During Hemodialysis (Regimen A)
Number analyzed (Participants) | 13 | 13
ug/mL | 70.5 [35.8 to 104] | 100 [56.5 to 211]

3. Other Pre Specified Outcome: Time to Maximum Concentration
Description: Sampling time at which maximum plasma concentration occurred, obtained directly from the experimental plasma concentration time data, without interpolation.
Time Frame: Up to 68 hours post dose
Measure: Median (Full Range); unit: Hours
Arm/Group | 6 mg/kg After Hemodialysis (Regimen B) | 9 mg/kg During Hemodialysis (Regimen A)
Number analyzed (Participants) | 13 | 13
Hours | 0.50 [0.50 to 1.00] | 0.50 [0.50 to 0.65]

4. Other Pre Specified Outcome: Half-life
Description: Apparent terminal half-life.
Time Frame: Up to 68 hours post dose
Measure: Median (Full Range); unit: Hours
Arm/Group | 6 mg/kg After Hemodialysis (Regimen B) | 9 mg/kg During Hemodialysis (Regimen A)
Number analyzed (Participants) | 13 | 13
Hours | 29.8 [19.7 to 38.1] | 31.1 [21.9 to 45.3]

5. Other Pre Specified Outcome: Clearance of Daptomycin
Description: Plasma clearance is dose (µg) divided by area under the concentration versus time curve from time 0 to last quantifiable concentration time.
Time Frame: Up to 68 hours post dose
Population: PK Population - defined as all subjects who received both doses of daptomycin
Measure: Median (Full Range); unit: mL/hr/kg
Arm/Group | 6 mg/kg After Hemodialysis (Regimen B) | 9 mg/kg During Hemodialysis (Regimen A)
Number analyzed (Participants) | 13 | 13
mL/hr/kg | 3.54 [2.38 to 6.23] | 3.32 [2.24 to 5.23]

6. Other Pre Specified Outcome: Volume of Distribution
Description: Volume of distribution at steady state (mL) calculated as the product of clearance and mean residence time.
Time Frame: Up to 68 hours post dose
Measure: Median (Full Range); unit: mL/kg
Arm/Group | 6 mg/kg After Hemodialysis (Regimen B) | 9 mg/kg During Hemodialysis (Regimen A)
Number analyzed (Participants) | 13 | 13
mL/kg | 137 [107 to 221] | 145 [115 to 219]

7. Secondary Outcome: Treatment-emergent Adverse Events
Description: Safety was monitored throughout the study, including observation and reports of AEs as well as changes in physical findings, vital signs, ECGs, and laboratory tests.
Time Frame: Up to 9 days after the last dose of study drug administration (Day 13 to Day 17 for those dosed on Day 8 and Day 20 to Day 24 for those dosed on Day 15).
Population: Safety population, defined as all subjects who received at least one dose of daptomycin
Measure: Number; unit: participants
Arm/Group | 6 mg/kg After Hemodialysis (Regimen B) | 9 mg/kg During Hemodialysis (Regimen A)
Number analyzed (Participants) | 15 | 13
participants | 2 | 3

ADVERSE EVENTS:
Time Frame: Up to 9 days after the last dose of study drug administration (Day 13 to Day 17 for those dosed on Day 8 and Day 20 to Day 24 for those dosed on Day 15).
Description: Safety was monitored throughout the study, including observation and reports of AEs as well as changes in physical findings, vital signs, ECGs, and laboratory tests.
Arm/Group | Sequence BA | Sequence AB
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 1/8 | 3/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sequence BA (N=8) | Sequence AB (N=7)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (2)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication is initiated by Cubist. If First Publication not published within 1 year of Study conclusion or termination, Investigator has right to publish and disclose the Data. Prior to any submission for publication, presentation, or communication of results or information arising from the Study, Investigator shall provide Cubist at least 90 days for review and comment upon the manuscript or other material for such publication or presentation.